CLINICAL TRIAL: NCT06375174
Title: SWISS-PRECISE (PERFUSION IMAGING TO IDENTIFY POSTERIOR CIRCULATION CANDIDATES FOR THROMBECTOMY)
Brief Title: PRECISE (PERFUSION IMAGING TO IDENTIFY POSTERIOR CIRCULATION CANDIDATES FOR THROMBECTOMY)
Acronym: SWISS-PRECISE
Status: Active, not recruiting | Type: Observational
Sponsor: Dr. med. Carlo Cereda (Other Government)
Responsible Party: Sponsor-Investigator, Dr. med. Carlo Cereda, PD Dr med., Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Other Study IDs: NSISTRCR_2202
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Posterior Circulation Acute Ischemic Stroke Due to Large Vessel Occlusion of the Vertebral or Basilar Artery Needing Endovascular Thrombectomy
MeSH Terms: interventions — Thrombectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thrombectomy — All procedures correspond to standard care and clinical routine

SUMMARY:
We hypothesize that patients with a favorable Critical Area Perfusion Score (CAPS≤3) on cerebral perfusion imaging will have a favorable response to revascularization by thrombectomy and that patients with a CAPS>3 will not

DETAILED DESCRIPTION:
PRECISE is a multicenter, prospective, observational cohort study. SWISS-PRECISE is a Switzerland Based spin-off of PRECISE with the intention to perform a final pooled analysis of data.

All procedures correspond to standard care and clinical routine. Perfusion imaging will be acquired prior to thrombectomy treatment. Enrolled patients have undergone standard of care baseline imaging with CT or MRI that includes angiography and cerebral perfusion imaging; therefore will be performed a control-MRI (or CT scan) after 24 hours and/or within 5±1 days from the thrombectomy, or before discharge.

Study procedures include the standard of care clinical follow-up assessments at uniform time intervals (5±1 days or discharge, 30±7 days, and 90±14 days). Data that will be collected on participants include: (1) all brain imaging; (2) demographics; (3) limited history; (4) blood pressure and vital signs before, during and after thrombectomy treatment; (5) NIHSS before and after thrombectomy treatment, at hospital discharge and at days 30 and 90 (if conducted in person); (6) discharge disposition; (7) modified Rankin Scale score prior to stroke, at discharge, and at days 30 and 90 (mRS will be assessed either in person or by phone); and (8) Quality of Life Assessment at day 90.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signs and symptoms consistent with an acute posterior circulation ischemic stroke 2. Baseline modified Rankin Scale (mRS) score ≤2 prior to qualifying stroke 3. Subjects age is 18-89 years, 90 or more if fully independent 4. Baseline National Institutes of Health Stroke Scale Score >4 and remains >4 immediately prior to thrombectomy treatment 5. Stroke symptoms began within 48 hours of thrombectomy treatment. Stroke onset is defined as the time the patient was last known to be at his/her neurologic baseline. Wake-up strokes are eligible if they meet the above time limits.

  6. Endovascular thrombectomy for BAO or PC-LVO planned as standard-of-care therapy (included aspiration, thrombectomy, angioplasty, stent placement, intravenous intrarterial GPIIb-IIIa inhibitor infusion) 7. Time of arterial puncture (femoral or radial artery) occurred (or expected to occur) within 120 minutes of CT or MR imaging study completion 8. Patient or Legally Authorized Representative has signed the study Informed Consent form

Exclusion Criteria:

* 1. Symptomatic stroke in another vascular territory (ie - MCA or ACA) 2. Other serious, advanced, or terminal illness (investigator judgment) or life expectancy is less than 6 months 3. Pre-existing medical, neurological, or psychiatric disease that would confound the neurological or functional outcomes evaluation 4. Any condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject Imaging

  1. Acute symptomatic arterial occlusions in more than one vascular territory on CTA (ie - associated anterior circulation LVO of the internal, middle, or anterior cerebral artery).
  2. Evidence of intracranial tumor (except small meningioma), acute intracranial hemorrhage, neoplasm or arteriovenous malformation
  3. Mass effect with significant herniation above the cerebral tentorium or below the foramen magnum
  4. Intracranial stent implanted in the same vascular territory that precludes safe deployment/removal of neurothrombectomy device.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Posterior circulation acute ischemic stroke due to large vessel occlusion of the vertebral or basilar artery needing endovascular thrombectomy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
mRS score | 5±1 days or discharge, 30±7 days, and 90±14 days
  Ordinal distribution of modified Rankin Scale (mRS) Scores 90 days after thrombectomy treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Neurocenter of Southern Switzerland, Ospedale Civico, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No